CLINICAL TRIAL: NCT00705302
Title: A Randomised Controlled Trial of the Effect of a Patient Education Program for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Patient Education in Patients With Chronic Obstructive Pulmonary Disease (COPD) - Effect and Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10307300; 17732 (Other: NSD); 4.2007.2589 (Other: REK)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; Outpatient; Patient education; Pulmonary rehabilitation; Self-management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Self-Help Groups; Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient education including self-help (Experimental): Patients in the arm will participate in a three months patient education and exercise program including a self-help group in 3 months of time.
  Interventions: Behavioral: Group training with self-help group
- patient education (Active Comparator): Patients in arm 2 will participate in the same patient education and exercise program as arm 1, but without an additional self-help group.
  Interventions: Behavioral: Group training

INTERVENTIONS:
Behavioral: Group training with self-help group — Combined educational and exercise program for pulmonary rehabilitation, with (1) or without(2 a self-help group. The educational part consists firstly of two days with group meetings with information from medical doctor, pharmacist, psychologist, ergonomist, nurse, social worker, physiotherapist and a clinical nutritional physiologist. One more day will be held after 3 months and it is the participants themselves who decide on the content of these days. An experienced patient will participate throughout the course. The exercise part consists of group training twice a week for 3 months with 10-15 participants in each group. Patients will instead of five of the group training sessions, participate in a self-help group.
  Arms: patient education including self-help
Behavioral: Group training — Combined educational and exercise program for pulmonary rehabilitation. The educational part consists firstly of two days with group meetings with information from medical doctor, pharmacist, psychologist, ergonomist, nurse, social worker, physiotherapist and a clinical nutritional physiologist. One more day will be held after 3 months and it is the participants themselves who decide on the content of these days. An experienced patient will participate throughout the course. The exercise part consists of group training twice a week for 3 months with 10-15 participants in each group.
  Arms: patient education

SUMMARY:
The aim of this study is to determine the long term effect of a self-help group in a patient education program for patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Pulmonary rehabilitation is aimed to increase the level of health of patients with COPD by increasing their self care ability. A recent updated systematic review concluded that evidence strongly supports respiratory rehabilitation as part of the spectrum of management of patients with chronic obstructive pulmonary disease (COPD). Studies of pulmonary rehabilitation programs lasting up to 18 months show that effects are mainly maintained throughout the duration of the program. The long term effect, however, is mostly studied for programs of shorter durations. Some of the studies with shorter duration have found that the achieved benefit was lost or diminished during the follow up period, while others have found that the effect has been maintained up to 18 months. Our necessity in the rehabilitative field is to find strategies to maintain benefits during time.

ELIGIBILITY:
Inclusion Criteria:

* (FEV1) lower that 75% of predicted
* the ability to participate in physical activity
* not been hospitalized the last month.

Exclusion Criteria:

* contraindications for physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) - Total score | Baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
Modified Borg scale (MBS) pre, during and post 6MWT | Baseline, 3, 6 and 12 months
Patient Activation Measure (PAM) | Baseline, 3, 6 and 12 months
The Perceived Quality of Life Scale | Baseline, 3, 6 and 12 months
6 minute walk test (6MWT) | Baseline, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, PhD, Study Director — Norwegian University of Technology and Science
Locations (1):
- Department of Public Health and General Practice, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Lomundal BK, Steinsbekk A. Observational studies of a one year self-management program and a two year pulmonary rehabilitation program in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2007;2(4):617-24. PMID 18268936
- [Background] Lomundal BK, Steinsbekk A. Five-year follow-up of a one-year self-management program for patients with COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:87-93. doi: 10.2147/COPD.S27352. Epub 2012 Feb 9. PMID 22371649